CLINICAL TRIAL: NCT01810146
Title: Characterization of the Digestive Functions and the Enteric Nervous System in Obesity. Investigations of Relationships With Metabolism Disorders(EnteroNeurObesity)
Brief Title: Characterization of the Digestive Functions and the Enteric Nervous System in Obesity. Investigations of Relationships With Metabolism Disorders (EnteroNeurObesity)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC12_0022
Record Dates: First submitted 2013-01-07; First posted 2013-03-13 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Obesity
Keywords: Patients eligible for bariatric surgery (BMI>40kg/m2)
MeSH Terms: conditions — Obesity

ARMS (1):
- Digestive functions investigations (No Intervention): Results from digestive functions investigations will be compared between patients eligible for bariatric surgery (BMI>40kg/m2) and volunteers (BMI between 20 and 25kg/m2).
  Interventions: Other: Digestive functions investigations

INTERVENTIONS:
Other: Digestive functions investigations

SUMMARY:
60 patients scheduled for bariatric surgery will be included into 3 categories (20 patients with non complicated obesity, 20 patients with metabolic syndrome and 20 patients with a type 2 diabetes or hypertension). 20 volunteers will be enrolled as normal referents. The patients and the volunteers will have a classical pre-operative check-up (fibroscopy, oesophageal pHmetry and manometry) and extra investigations as isotopic gastric empty exam, lactulose oro-caecal transit exam, intestinal permeability test calculated by lactulose-manitol ratio urinary excretion. Intestinal and colonic biopsies will be also provided for studying permeability. For only patients, samples from the gastric resection will be provided for analysing the enteric nervous system and motricity.

ELIGIBILITY:
Patients:

Patients must be aged between 18 and 65 years old with a BMI>40kg/m2 for non complicated patients or with a metabolic syndrome and with a BMI>35kg/m2 for patients with type 2 diabetes or hypertension. They must be eligible for bariatric surgery.

Patients with a type 1 diabetes, neurologic or neuro-degenerative disease will be excluded.

Volunteers:

Volunteers must be aged between 18 and 65 years old with a BMI between 20 and 25kg/m2 Men and women are eligible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
T1/2 solids (on the kinetic of isotopic gastric empty exam) | 6 months
  This evaluation will be obtained before bariatric surgery for patients and at any time before end of study for volunteers.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, France